CLINICAL TRIAL: NCT04120805
Title: Randomized, Prospective Evaluation of Hemostatic Agents in Robotic-Assisted Laparoscopic Partial Nephrectomy
Brief Title: Random Evaluation of Patients Who Have Had Laparoscopic Partial Nephrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB15-0519
Record Dates: First submitted 2019-01-14; First posted 2019-10-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (Hemostatic Agents Plus +) (Experimental)
  Interventions: Device: Hemostatic Agent
- Group 2 (Hemostatic Agents Negative -) (Active Comparator): No Hemostatic Agent
  Interventions: Other: No Hemostatic Agent

INTERVENTIONS:
Device: Hemostatic Agent — Patients undergoing robotic-assisted laparoscopic partial nephrectomy with the use of hemostatic agents by a surgeon
  Arms: Group 1 (Hemostatic Agents Plus +)
Other: No Hemostatic Agent — Patients undergoing robotic-assisted laparoscopic partial nephrectomy without the use of hemostatic agents by a surgeon
  Arms: Group 2 (Hemostatic Agents Negative -)

SUMMARY:
The purpose of this study is to evaluate the necessity of using hemostatic agents as a tool when performing robotic partial nephrectomy in the treatment of kidney cancer. This project asks whether patients who undergo robotic partial nephrectomy without the surgeon using hemostatic agents during the procedure will have the same, fewer, or more complications than when patients undergo this same surgery with the surgeon using hemostatic agents during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years and older.
2. Patients must have a solid or cystic renal mass suspicious for malignancy by imaging with ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI).
3. Patients must be initially scheduled RALPN as opposed to radical nephrectomy or other techniques for partial nephrectomy such as open surgery or pure laparoscopy without robot assistance.
4. Patients with bilateral kidneys or a solitary kidney, so long as these are native kidneys as opposed to a transplanted kidney.
5. Patients can have the common single renal artery and single renal vein, or they can have common variants such as two renal arteries and/or two renal veins.

Exclusion Criteria:

1. Patients on hemodialysis.
2. Patients who have had a renal transplantation.
3. Patients on therapeutic anticoagulation prior to surgery (example anticoagulants include: aspirin 325 mg daily, clopidogrel, warfarin, fondaparinux, dabigatran, and rivaroxaban). However, patients who take aspirin 81 mg daily as their daily regimen will be included.
4. Patients with bleeding disorders (example: hemophilia) and other documented coagulopathy (example: chronic liver disease) with INR greater than 1.0 at baseline.
5. Patients who have had a prior surgical procedure, aside from percutaneous renal biopsy, on the kidney in the current operation.
6. Patients with over 100 mL of estimated blood loss (calculated by anesthesia team using the suction canisters) prior to clamping of the renal hilum will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
An absolute change in hemoglobin | up to 6 months
  The change in hemoglobin will be measured as the difference between the hemoglobin obtained postoperatively and the hemoglobin obtained preoperatively.

SECONDARY OUTCOMES:
Total number of major bleeding complications | up to 6 months
  Major complications are blood loss requiring transfusion of packed red blood cells, reoperation and endovascular ablation
Safety monitoring parameters: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 6 months
  Safety monitoring parameters including stroke, death, cardiac arrest, myocardial infarction and urine leak
Operating room parameters | up to 6 months
  Operating room parameters including number of sutures used during renorrhaphy and capsular closure, duration of renorrhaphy and patients in group 2 with no hemostatic agents who required HA at the surgeons discretion
Patients with a hospital stay over 30 days | up to 6 months
  Total length of all inpatient hospital stay over 30 days measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Shalhav, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States